CLINICAL TRIAL: NCT06109155
Title: The Dose Effect of Activated Clotting Time and Tranexamic Acid on Bleeding in Adult Cardiac Surgery
Brief Title: The Effect of ACT and Tranexamic Acid on Bleeding in Cardiac Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF23323A
Record Dates: First submitted 2023-09-22; First posted 2023-10-31 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Surgery, Cardiac; Tranxemic Acid; Activated Clotting Time; Heparin; Cardiopulmonary Bypass
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: During cardiac surgery with cardiopulmonary bypass support, participants will be divided into 4 groups. During procedure, they will recieve different doses of tranexamic acid and different level of activated clotting time. Then, we will monitor the amount of blood loss and blood transfusion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the research process, any raw data will be kept and encrypted by the principal investigator, and it will not be accessible or interpretable by others.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- High dose tranexamic acid + high ACT level (Active Comparator): high dose tranexamic acid: 50mg/kg ACT level: > 600 sec
  Interventions: Drug: Tranexamic acid
- High dose tranexamic acid + low ACT level (Active Comparator): high dose tranexamic acid: 50mg/kg ACT level: 400~ 600 sec
  Interventions: Drug: Tranexamic acid
- Low dose tranexamic acid + low ACT level (Active Comparator): Low dose tranxeamic acid: 20mg/kg ACT level: 400~ 600 sec
  Interventions: Drug: Tranexamic acid
- Low dose tranexamic acid + high ACT level (Placebo Comparator): Low dose tranxeamic acid: 20mg/kg ACT level: > 600 sec
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — tranexamic acid will be used in two different doses (50mg/kg vs 20mg/kg). the tranexamic acid pump will start from the begin of anesthesia until all dose is administrated.

SUMMARY:
The goal of this clinical trial is to the dose effect of tranexamic acid and the level of ACT on bleeding in adult cardiac surgery.

The main questions it aims to answer are:

1. Does higher dose of tranexamic acid reduce the amount of bleeding and blood transfusion?
2. Does lower ACT level during cardiac surgery reduce the amount of bleeding and blood transfusion?

Participants will divided into four groups which have different tranexamic acid dose and ACT level during cardiac surgery to see if there is any different in the amount of bleeding and blood transfusion.

DETAILED DESCRIPTION:
This study is going to analyze the medical records of patients who underwent cardiac surgery between December 1, 2023, and December 31, 2026.

The investigators will categorize patients into four groups based on anticoagulation indices (ACT 400-600 seconds; ACT > 600 seconds) and tranexamic acid dosages (low dose; high dose) within the range considered safe for CPB.

The primary outcome will be the volume of postoperative bleeding within 24 hours for each group.

The findings of this study will contribute to the existing clinical evidence and provide insights for the monitoring and pharmacological management in cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult, cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* pregnant
* emergency procedure
* immune compromised
* aortic surgery
* end-stage renal disease
* liver disease
* critical status
* incomplete clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood loss | 24 hours
  monitor the amount of blood loss after procedure
blood transfusion | procedure time, an average of 6 hours
  the amount of blood transfusion during procedure

SECONDARY OUTCOMES:
30-day mortality | 30 days
  30-day mortality after procedure

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Taichung Veterans General hospital, Taichung

IPD SHARING:
Plan to Share IPD: No